CLINICAL TRIAL: NCT00893893
Title: Very-low-density-lipoprotein Triglyceride(VLDL-TG) Uptake in Visceral Fat
Brief Title: Very-low-density-lipoprotein Triglyceride (VLDL-TG) Uptake in Visceral Fat
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Esben Søndergaard, MD, ph.d., University of Aarhus
Other Study IDs: ES-0003
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Healthy; Obesity
Keywords: Obesity; Lipid metabolism; VLDL
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Adipose tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Lean premenopausal women
- 2: Visceral obese premenopausal women

SUMMARY:
Purpose:

To investigate the uptake of VLDL-TG in visceral fat in lean and overweight individuals

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age: 20-50 years
* Premenopausal

Exclusion Criteria:

* Smoking
* Alcohol abuse
* Use of medications

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology M, Aarhus Hospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Sondergaard E, Nellemann B, Sorensen LP, Gormsen LC, Christiansen JS, Ernst E, Dueholm M, Nielsen S. Similar VLDL-TG storage in visceral and subcutaneous fat in obese and lean women. Diabetes. 2011 Nov;60(11):2787-91. doi: 10.2337/db11-0604. Epub 2011 Sep 12. PMID 21911742